CLINICAL TRIAL: NCT03895216
Title: Identification and Characterization of Predictive Factors of Onset of Bone Metastases in Cancer Patients
Acronym: PreMetOn
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Gianluca Giavaresi, MD, MD, Istituto Ortopedico Rizzoli
Other Study IDs: CE AVEC 352/2018/Sper/IOR
Record Dates: First submitted 2019-03-22; First posted 2019-03-29 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Bone Metastases
Keywords: MicroRNAs; Bone Metastases; Exosomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma and circulating exosomes, microRNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the present study is to identify deregulated miRNAs in oncological patients with bone metastases present within the circulating exosomes and responsible for the biological mechanisms involved in the process of bone metastasis, in order to obtain a panel of biomarkers predictive of this risk.

Through appropriate molecular screening methods a specific panel of significantly deregulated miRNAs will be identified; subsequently bioinformatics analyzes through the use of dedicated databases will be carried out, based on literature data and predicted protein targets in order to identify their potential role in tumor progression, and especially in the onset of bone metastases. Attention, therefore, may be focused on the individual miRNAs identified through individual analysis analyzes of gene expression. These biomarkers could also serve as therapeutic targets, allowing to improve the effectiveness of current therapies and to undertake timely and appropriate therapeutic choices, developed on the basis of the patient's molecular characteristics

DETAILED DESCRIPTION:
MATERIALS AND METHODS: 1) Removal of whole blood from peripheral vein and separation of plasma from enrolled metastatic cancer patients; 2) Isolation of tumor exosomes circulating from the plasma of cancer patients (Kit Invitrogen: Total Exosome Isolation Reagent); 3) Next generation sequencing methods (NGS) will be used to evaluate the expression profiles of miRNAs isolated from circulating tumor exosomes (MiSeq Illumina System); 4) Mass spectrometry methods will be used for the proteome analysis of circulating exosomes isolated from the plasma of cancer patients (Triple TOFF 5600 Plus System AND HPLC analysis of bioactive and biomarker peptides); 5) 3D cultures for the study of cross-talk between circulating tumor exosomes (isolated from the patients' plasma) and bone tissue cells (using commercial cell lines) as part of the metastatic process (Cellec perfusion bioreactor BioteK AG).

Enrollment Procedures: Patients considered eligible will be enrolled in the study, after providing a written informed consent.

Data Collection: Clinical data will be retrieved by patient's source document. A protocol-specific CRF reporting the results of the analyses will be provided. A CRF is required and should be completed for each included subject.

Ethics: The clinical trial protocol and its documents will be sent before initiating the study to the competent Authorities and Ethics Committees of each participating country for its approval. The responsible investigator will ensure that this study is conducted in agreement with either the most updated Declaration of Helsinki and all the international and local laws that apply to clinical trials and to patient protection. The protocol has been written, and the study will be conducted according to the principles of the ICH Harmonized Tripartite Guideline for Good Clinical Practice (ref: http://www.emea.eu.int/pdfs/human/ich/013595en.pdf).

Informed Consent: All patients will be informed, by the investigator, of the aims of the study, the possible risks and benefits that will derive from the study participation. The Investigator must clearly inform that the patient is free to refuse participation in the study and that can withdraw consent at any time and for any reason. They will be informed as to the strict confidentiality of their patient data, but that their medical records may be reviewed for trial purposes by authorized individuals other than their treating physician. The informed consent procedure must conform to the ICH guidelines on Good Clinical Practice. This implies that "the written informed consent form should be signed and personally dated by the patient or by the patient's legally acceptable representative".

The Investigator must also sign the Informed Consent form, and will keep the original at the site and a copy of the original must be handed to the patient.

The competent ethics committee for each Institution participating to the study must validate local informed consent documents before the study can be opened. It will be emphasized that the participation is voluntary and that the patient is allowed to refuse further participation in the study whenever he/she wants. This will not prejudice the patient's subsequent care.

General Principles for Human Biological Material (HBM) collection: Human biological material (HBM) collection involves the collection and storage of biological material, residual biological material or derivatives in compliance with ethical and technical requirements. Biological material (blood samples) will be centralized and stored at Istituto Ortopedico Rizzoli - Dipartimento Rizzoli-Sicilia, Bagheria (Palermo). From here, the biological material will be used and stored according with the sample characteristic and applicable regulation.

Plasma and circulating exosomes obtained from blood will be stored inside sterile containers (falcon, tubes, eppendorf) in a freezer at the temperature of -80 °C at the Istituto Ortopedico Rizzoli -Dipartimento Rizzoli Sicilia.

The following principles apply to storage of HBM: (a) The Istituto Ortopedico Rizzoli will have a designated person responsible for collection and will act as a communication point; (b) The collected HBM should be documented, i.e. the amount remaining and its location. act as a communication point; and (c) The storage and use of biological material will take place in accordance with the standards of good laboratory practice (GLP) and applicable legislation.

Confidentiality: In order to ensure confidentiality of clinical trial data as disposed the national and European applicable regulation, data will be only accessible for the trial Sponsor and its designees, for monitoring/auditing procedures, the Investigator and collaborators, the Ethics Committee of each corresponding site and the Health Authority. Investigator and the Institution will allow access to data and source documentation for monitoring, auditing, Ethic Committee revision and inspections of Health Authority, but maintaining at all times subject personal data confidentiality as specified in the applicable regulation.

The Investigator must guarantee that patient anonymity is kept at all times and their identity must be protected from unauthorized persons and institutions.

All patients included in the study will be identified with a numeric code, so that no identifiable personal data will be collected. The Investigator must have and conserve a patients' inclusion registry where it figures the personal data of the patient: name, surname, address and corresponding identification code into the study, this register will be kept on the Investigator File.

Publication policy and data ownership: The principal investigator of the study is responsible for the final report, of the publication publish all the data collected as described in the protocol and will ensure that the data are reported responsibly and consistently. In particular, the publication of data deriving from the present study will take place independently of the results obtained. The transmission or dissemination of data, through scientific publications and / or presentation at conferences, congresses and seminars, will take place exclusively following the purely statistical processing of the same, or in an absolutely anonymous form. All the study data are owned by the sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of oncological pathology with evidence of disease progression and presence of bone metastases;
* Patients who have to undergo biopsy of bone metastases or clinical metastasectomy. The analysis of the circulated biomarkers is done in all patients who are subjected to biopsy or metastasis resection to be sure of the diagnosis of bone metastasis, and to have the opportunity to follow patients in the follow-up provided by this type of surgical treatment.
* Life expectancy over 6 months;
* Patients able to provide written informed consent to the study.

Exclusion Criteria:

* Severe cognitive deficits or psychiatric disorders;
* Patients who do not wish or cannot comply with the study protocol;
* Women of childbearing age who are pregnant or breast-feeding. The protocol excludes pregnant patients because, in the case of metastasectomy, the anesthesia associated with this procedure is completely discouraged in pregnant women and, in addition, any factor is to be avoided (such as a different hormonal arrangement linked to pregnancy ) that can jeopardize or introduce a bias in the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A maximum number of 25 patients with metastatic bone lesions is expected to be enrolled and who must undergo metastasectomy or who must perform a bone biopsy of the metastasis. Patients will be enrolled in the clinical trial only after providing written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in miRNAs content of circulating tumor exosomes | Within 24 hours before surgery, within 48 hours of metastasectomy or bone biopsy, and follow-up checks at 1, 3, 6 months and 1 year
  Identification of miRNA isolated from circulating tumor exosomes and their changes will be done through expression profiling studies using Next Generation Sequencing (NGS) during follow-up time points. Molecular characterization will be performed on miRNA samples isolated from circulating tumor exosomes separated from the plasma in order to identify new markers related to tumor progression (bone metastases).
Change in protein content of circulating tumor exosomes | Within 24 hours before surgery, within 48 hours of metastasectomy or bone biopsy, and follow-up checks at 1, 3, 6 months and 1 year
  Qualitative and quantitative proteomic analysis of the content of circulating tumor exosomes will be performed by using Triple TOF mass spectrophotometer and variation during follow-up time points wil be measured.

SECONDARY OUTCOMES:
Relationship between plasma levels of circulating tumor exosomes and their content in miRNAs with overall survival and progression of the disease. | Within 24 hours before surgery, within 48 hours of metastasectomy or bone biopsy, and follow-up checks at 1, 3, 6 months and 1 year
  Correlation analyses (correlation coefficients) among plasma levels of circulating tumor exosomes, their content in miRNAs, and clinical parameters related to patient survival and progression of their disease.
Cross-talk between isolated circulating tumor exosomes and commercial lines of bone tissue cells in the metastatic process. | Within 24 hours before surgery, within 48 hours of metastasectomy or bone biopsy, and follow-up checks at 1, 3, 6 months and 1 year
  In vitro studies with 3D culture model will then allow a more detailed understanding of the cross-talk between tumor exosomes and bone tissue cells (commercial cell lines) within the tumor niche.

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Giavaresi, MD, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Dipartimento Rizzoli Sicialia - Istituto Ortopedico Rizzoli, Bagheria, Palermo, Italy

REFERENCES:
- [Result] Raimondi L, De Luca A, Costa V, Amodio N, Carina V, Bellavia D, Tassone P, Pagani S, Fini M, Alessandro R, Giavaresi G. Circulating biomarkers in osteosarcoma: new translational tools for diagnosis and treatment. Oncotarget. 2017 Aug 3;8(59):100831-100851. doi: 10.18632/oncotarget.19852. eCollection 2017 Nov 21. PMID 29246026
- [Result] Graveel CR, Calderone HM, Westerhuis JJ, Winn ME, Sempere LF. Critical analysis of the potential for microRNA biomarkers in breast cancer management. Breast Cancer (Dove Med Press). 2015 Feb 23;7:59-79. doi: 10.2147/BCTT.S43799. eCollection 2015. PMID 25759599
- [Result] Macias M, Alegre E, Diaz-Lagares A, Patino A, Perez-Gracia JL, Sanmamed M, Lopez-Lopez R, Varo N, Gonzalez A. Liquid Biopsy: From Basic Research to Clinical Practice. Adv Clin Chem. 2018;83:73-119. doi: 10.1016/bs.acc.2017.10.003. Epub 2017 Nov 23. PMID 29304904
- [Result] Kai K, Dittmar RL, Sen S. Secretory microRNAs as biomarkers of cancer. Semin Cell Dev Biol. 2018 Jun;78:22-36. doi: 10.1016/j.semcdb.2017.12.011. Epub 2017 Dec 19. PMID 29258963
- [Result] Li A, Zhang T, Zheng M, Liu Y, Chen Z. Exosomal proteins as potential markers of tumor diagnosis. J Hematol Oncol. 2017 Dec 27;10(1):175. doi: 10.1186/s13045-017-0542-8. PMID 29282096